CLINICAL TRIAL: NCT01452932
Title: Muscle Training Effectiveness in the Degree of Dyspnea and Aerobic Capacity in COPD in an Institution Health Service Provider in the Department of Antioquia
Brief Title: Muscle Training Effectiveness in the Degree of Dyspnea and Aerobic Capacity in COPD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CES University (Other)
Collaborators: La ceja Hospital (Unknown)
Responsible Party: Principal Investigator, Nathalia Suarez, Principal investigator, CES University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCESCOPD
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Dyspnea
Keywords: Chronic obstructive pulmonary disease; Dyspnea; Exercise test; Endurance training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Physical Therapy Modalities; Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy (Experimental): Group of participants who recive physiotherapy treatment using Kabat technique for the upper limbs resistance training during 12 weeks
  Interventions: Other: Physiotherapy
- Yoga (Other): Group of participants who recive Yoga sessions during 12 weeks
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Physiotherapy — The physiotherapeutic intervention was based on the Kabat (PNF) technique. Thirty-three sessions were planed. Each session lasted between thirty and fifty minutes.
  The experimental group was guided by a physiotherapist or a physiotherapy student and each session took place in a hospital auditorium provided with oxygen cylinders, chairs and water.
  Each session consisted of a warm up and stretch period, a period of resistance training of the upper limbs with their rest periods in which diaphragmatic breathing exercises and finally a cooling period.
  The instructions and instruments given to each participant such as weights and elastic bands were the same for all of them.
  Arms: Physiotherapy
Other: Yoga — The intervention for the other group was the Yoga technique. Thirty-six sessions were planed. Each session was based on breathing, relaxation, and stretching exercises. Each session lasted between thirthy and forty minutes.
  The group was led by a Yoga Instructor and each sessions took place in a hospital auditorium provided by oxygen cylinders, chairs and water.
  No instruments were needed for this intervention.
  Arms: Yoga

SUMMARY:
Objective: To estimate the effectiveness of muscle training, the degree of dyspnea and aerobic capacity in patients over 50 with COPD, in a health care institution provider in Antioquia.

Question: What is the effectiveness of muscle training, in the degree of dyspnea and aerobic capacity in COPD patients over 50 years, in a health service institution provider in the department of Antioquia?

Hypothesis: Muscle training causes changes in the degree of dyspnea and aerobic capacity, other than the breathing exercises and relaxation

Design: Randomized clinical trial with allocation and blinding of the autcomes assesor.

Participants: COPD patients stage II and II, male and female, over 50 years old, who are attending to a community health service provider in the department of Antioquia.

Intervention: A physiotherapeutic intervention using PNF technique was applied to the experimental physiotherapy group versus Yoga sessions applied to the other group. Twelve weeks protocol performing three sessions per week.

Outcome measures: Dyspnea degree and aerobic capacity was measured using the MMRC scale and the six minute walking test respectively at the begining and the end of the study.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is defined by GOLD (The Global Initiative for Chronic Obstructive Lung Disease) as a disease process characterized by progressive airflow limitation associated with an abnormal inflammatory response of the lungs to particles or harmful gases and is not fully reversible. This restriction generates an expiratory flow of air entrapment resulting hyperinflation, coupled with the effects that systemic, structural changes occur in skeletal muscles which leads to greater fatigue causing dyspnea. Consequently, patients with COPD require participation of accessory muscles of respiration, which should have a dual function during activities involving the upper limbs, to supply the ventilatory requirements and movements of the shoulder girdle, which increases dyspnea carrying the patient to stop their activities, leading to physical deconditioning and progressively decreasing aerobic capacity. This demonstrates the need to improve the resistance of the upper limb muscles in these patients, thus contributing to a reduction in the degree of dyspnea and improved their aerobic capacity. The investigators propose a study aimed at determining the effectiveness of muscle training in the degree of dyspnea and aerobic capacity in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 50 years with a diagnosis of COPD stage II and III according to GOLD classification, performed spirometry
* Patients who manifest dyspnea on MRC
* Patients SGSS affiliates.
* COPD controlled, verified medical history
* Voluntary participation in informed consent

Exclusion Criteria:

* Higher mental functions altered
* Degenerative musculoskeletal diseases (acute state)
* Multisystem disease not controlled
* Perform a current fitness program

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Dyspnea degree | Up to 12 weeks
  The degree of dyspnea is measured at baseline as one of the most important criteria for inclusion, after randomization of participants and past twelve weeks (duration of the intervention protocol) is measured this variable as a primary outcome.
Aerobic capacity | Up to 12 weeks
  Aerobic capacity is measured with the six minutes walking test (6MWT) at baseline as one of the most important criteria for inclusion, performed after randomization of participants and past twelve weeks (duration of the intervention protocol) is measured this variable as a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalia Suarez, Profesional, Principal Investigator — Professor CES University